CLINICAL TRIAL: NCT02303587
Title: Low Dose Versus High Dose Methylprednisolone for Children With Severe Mycoplasma Pneumoniae Pneumonia : a Multicenter Randomized Blinded Trial
Brief Title: Methylprednisolone for Children With Severe Mycoplasma Pneumoniae Pneumonia (MCMP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Children's Hospital (Other)
Collaborators: Shengjing Hospital (Other); Children's Hospital of The Capital Institute of Pediatrics (Other); Shanxi Provincial Maternity and Children's Hospital (Other); Baoding Children's Hospital (Other)
Responsible Party: Principal Investigator, Baoping XU, Chief of Respiratory Department, Beijing Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BCHlung001
Record Dates: First submitted 2014-11-21; First posted 2014-12-01 (Estimated); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Mycoplasma Pneumoniae Pneumonia
Keywords: Severe mycoplasma pneumoniae; pneumonia; children
MeSH Terms: conditions — Pneumonia, Mycoplasma; Pneumonia | interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- low dose group (Experimental): methylprednisolone 2mg-4mg/Kg
  Interventions: Drug: methylprednisolone
- high dose group (Experimental): methylprednisolone 10mg/Kg
  Interventions: Drug: methylprednisolone

INTERVENTIONS:
Drug: methylprednisolone

SUMMARY:
The study is designed to investigate difference in percentage of presentation of atelectasis, bronchiectasis, bronchiolitis obliterans, or consolidation in 6 months after discharge in those treated with a low dose regimen of methylprednisolone initiated with 2 or 4 mg/kg/d for 3 days followed by tapering, combined with sequential treatment with azithromycin versus a high dose regimen of methylprednisolone initiated with 10 mg/kg/d for 3 days followed by tapering, combined with sequential treatment with azithromycin.

DETAILED DESCRIPTION:
Mycoplasma pneumonia pneumonia (MPP) accounts for approximately 10-30% of childhood community-acquired pneumonia (CAP) in China. Macrolide is the first choice for MPP. However, progression to severe pneumonia might occur despite antibiotics therapy. And some patients have sequelae of bronchiolitis obliterans, bronchiectasis and atelectasis, et al. Based on inflammatory and immunological mechanism, there is some clinical evidence that adjuvant of corticosteroid reduced morbidity and improved the outcome in the children with severe MPP. However, the dosage of corticosteroid varied greatly in studies. Therefore, a large prospective study is needed to define the benefits of high-dose corticosteroid therapy in MPP.

Patients will be randomized into two groups: the low dose group and the high dose group. The low dose group will receive methylprednisolone 2 or 4 mg/kg/d for 3 days followed by tapering in 9 days, combined with sequential treatment with azithromycin. The high dose group will receive methylprednisolone 10 mg/kg/d for 3 days followed by tapering in 9 days, combined with sequential treatment with azithromycin. After discharge, patients of both groups will be followed up at 1, 3, and 6 months.

The number of pulmonary lesions, including atelectasis, bronchiectasis, bronchiolitis obliterans, or consolidations, in 6 months after discharge will be compared in two groups. The number of adverse events, such as hyperglycemia, hypertension, increased intraocular pressure, will be compared between the two groups.

The trial will be completed in 36 months, with 424 subjects recruited from 5 hospitals in partnership with clinical research collaboration of National Clinical Research Center for Respiratory Diseases.

ELIGIBILITY:
Inclusion Criteria:

Severe pneumonia diagnosis criteria were based on the "Zhu Futang Practical Pediatrics" (the 7th Edition) and "the guideline of management of community-acquired pneumonia in children in China"(Chinese Journal of Pediatrics, 2013, 51:745-752, 856-862). Severe pneumonia is defined as pneumonia with one of the following:

1. Less than 18 years old
2. Severe pneumonia that is defined as pneumonia with one of the followings:

   * poor general condition
   * increased respiratory rate( infant>70/min，older children>50/min)
   * dyspnea
   * cyanosis
   * multilobe involvement or ≥ 2/3 lung involvement
   * extrapulmonary complication
   * pleural effusion
   * Transcutaneous oxygen saturation in room air ≤92%
3. Serum M. pneumoniae antibody≥ 1:320, or serum M. pneumoniae antibody≥ 1:160 with positive PCR of M. pneumoniae or seroconversion (increased antibody titers ≥4 folds) Subject/Guardian is informed and consent.

Exclusion Criteria:

Subject will be excluded if she or he has one of the following:

* evidence of bacterial pneumonia;
* evidence of viral pneumonia;
* evidence of fugal pneumonia;
* evidence of pulmonary tuberculosis;
* respiratory failure requiring mechanical ventilation;
* hemophagocytic syndrome;
* liver failure or renal insufficiency;
* congenital heart disease;
* heart failure;
* kidney disease;
* connective tissue disease;
* immunodeficiency;
* tumor;
* a history of hypertension or diabetes mellitus;
* recurrent respiratory tract infection;
* congenital bronchopulmonary dysplasia;
* increased intraocular pressure;
* history of use of glucocorticoids ≥1 week in previous 3 months;
* having contraindications to glucocorticoids or azithromycin;
* using of immunosuppressant before randomization;
* undergoing trial for other medications or instruments.

Ages: 29 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 424 (Actual)
Dates: Start 2014-12; Primary Completion 2019-10-16 (Actual); Study Completion 2019-10-16 (Actual)

PRIMARY OUTCOMES:
pulmonary lesions | 6 months
  Pulmonary lesions include atelectasis, bronchiectasia, bronchiolitis obliterans, consolidation

SECONDARY OUTCOMES:
recovery time of temperature | 2 weeks
the proportion of absorption of pulmonary lesions | 2 weeks
duration of hospitalization, | 2 weeks
number of participant(s ) need intensive care | 2 weeks
number of participant(s )with acute respiratory distress syndrome | 2 weeks
number of participant(s) with hemophagocytic syndrome | 2 weeks
number of participant(s) with hyperglycemia | 2 weeks
number of participant(s) with hypertension | 6 months
number of participant(s) who died during the trial | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kunling Shen, MD,PhD, Study Director — Beijing Children's Hospital of Capital Medical University, China; Baoping Xu, MD, PhD, Principal Investigator — Beijing Children's Hospital of Capital Medical University, China; Xiaoxia Peng, MD, PhD, Principal Investigator — Beijing Children's Hospital of Capital Medical University, China
Locations (1):
- Beijing Children's Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chinese maternal and child health development report (2011). The Ministry of health of the people's Republic of China
- [Background] Nagalingam NA, Adesiyun AA, Swanston WH, Bartholomew M. Prevalence of Mycoplasma pneumoniae and Chlamydia pneumoniae in pneumonia patients in four major hospitals in Trinidad. New Microbiol. 2004 Oct;27(4):345-51. PMID 15646048
- [Background] QIN Ming, TIAN Man, XIA Wen, ect. Etiology of community-acquired pneumonia in children.THE JOURNAL OF CLINICAL PEDIATRICS,2008,26(4):312-315.
- [Background] Eun BW, Kim NH, Choi EH, Lee HJ. Mycoplasma pneumoniae in Korean children: the epidemiology of pneumonia over an 18-year period. J Infect. 2008 May;56(5):326-31. doi: 10.1016/j.jinf.2008.02.018. Epub 2008 Apr 16. PMID 18420275
- [Background] Gaillat J, Flahault A, deBarbeyrac B, Orfila J, Portier H, Ducroix JP, Bebear C, Mayaud C. Community epidemiology of Chlamydia and Mycoplasma pneumoniae in LRTI in France over 29 months. Eur J Epidemiol. 2005;20(7):643-51. doi: 10.1007/s10654-005-5868-9. PMID 16119439
- [Background] YU Zhen-xi, LIU Xiu-yun, JIANG Zai-fang. Analysis of relevant factors of severe mycoplasma pneumoniae pneumonia in acute phase in children. JOURNAL OF APPLIED CLINICAL PEDIATRICS, 2011，26（4）：246-249.
- [Background] Zhang Q, Guo Z, Bai Z, MacDonald NE. A 4 year prospective study to determine risk factors for severe community acquired pneumonia in children in southern China. Pediatr Pulmonol. 2013 Apr;48(4):390-7. doi: 10.1002/ppul.22608. Epub 2012 Jul 6. PMID 22778084
- [Background] Hirao S, Wada H, Nakagaki K, Saraya T, Kurai D, Mikura S, Yasutake T, Higaki M, Yokoyama T, Ishii H, Nakata K, Aakashi T, Kamiya S, Goto H. Inflammation provoked by Mycoplasma pneumoniae extract: implications for combination treatment with clarithromycin and dexamethasone. FEMS Immunol Med Microbiol. 2011 Jul;62(2):182-9. doi: 10.1111/j.1574-695X.2011.00799.x. Epub 2011 Apr 11. PMID 21395697
- [Background] Shimizu T, Kida Y, Kuwano K. Cytoadherence-dependent induction of inflammatory responses by Mycoplasma pneumoniae. Immunology. 2011 May;133(1):51-61. doi: 10.1111/j.1365-2567.2011.03408.x. Epub 2011 Feb 14. PMID 21320122
- [Background] Tamura A, Matsubara K, Tanaka T, Nigami H, Yura K, Fukaya T. Methylprednisolone pulse therapy for refractory Mycoplasma pneumoniae pneumonia in children. J Infect. 2008 Sep;57(3):223-8. doi: 10.1016/j.jinf.2008.06.012. Epub 2008 Jul 25. PMID 18656264
- [Derived] Xu B, Peng X, Yao Y, Yin J, Chen L, Liu J, Wang H, Gao L, Shen A, Shen K. Low-dose versus high-dose methylprednisolone for children with severe Mycoplasma pneumoniae pneumonia (MCMP): Study protocol for a randomized controlled trial. Pediatr Investig. 2018 Oct 17;2(3):176-183. doi: 10.1002/ped4.12041. eCollection 2018 Sep. PMID 32851257